CLINICAL TRIAL: NCT01408927
Title: Prevalence and Level of Thienopyridine Resistance Seen in a Contemporary PCI and CABG Population
Brief Title: Prevalence and Level of Thienopyridine Resistance Seen in a Contemporary Percutaneous Coronary Intervention or Coronary Artery Bypass Graft Population
Acronym: VASP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: VASP
Record Dates: First submitted 2011-07-28; First posted 2011-08-03 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Increased Drug Resistance
Keywords: Thienopyridine resistance; Aspirin resistance; Platelet reactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Thienopyridine resistance testing — Thienopyridine resistance will be measured by flow cytometry of vasodilator-stimulated phosphoprotein (VASP) phosphorylation, and/or VerifyNow P2Y12 assay, and/or the Chrono-Log Lumi-Aggregometer, and/or the PlaCor PRT 7000 platelet reactivity assay.
Other: Aspirin resistance testing — Aspirin resistance will be measured by the VerifyNow aspirin resistance assay.
Other: Genetic polymorphism assessment — The presence of minor alleles in selected single nucleotide polymorphisms (SNPs) as measured by the Applied Biosystems Open Array system.

SUMMARY:
The primary objective of this prospective clinical registry is to determine the prevalence and level of thienopyridine resistance seen in a population undergoing contemporary percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG).

DETAILED DESCRIPTION:
This is a prospective cohort study of 1000 patients presenting to the Washington Hospital Center for percutaneous coronary intervention or coronary artery bypass surgery.

The aim of this prospective clinical registry is to determine the prevalence and level of thienopyridine resistance seen in a population presenting for cardiac catheterization and undergoing percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG). Thienopyridine resistance will be measured by flow cytometry of the vasodilator-stimulated phosphoprotein (VASP) phosphorylation, and/or the VerifyNow P2Y12 assay, and/or the Chrono-Log Lumi-Aggregometer, and/or the PlaCor PRT 7000 platelet reactivity assay.

A secondary objective of this study is to correlate a variety of genetic polymorphisms with levels of platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient >18 years old.
2. PCI group only: Patient scheduled to undergo cardiac catheterization or underwent percutaneous coronary intervention (PCI), during hospital stay.
3. CABG group only: Patient is scheduled to undergo, or has underwent, coronary artery bypass surgery with at least one saphenous vein graft.
4. Treated with a loading dose of clopidogrel or prasugrel at least 6 hours prior to the blood draw, or on a maintenance dose of clopidogrel or prasugrel for a minimum of 5 days.
5. Genetic testing subgroup only: Patient has undergone PCI (only), and has been treated with a thienopyridine as in 4.

Exclusion Criteria:

1. Known allergies to aspirin, clopidogrel, or prasugrel;
2. Use of a glycoprotein (GP) IIb/IIIa within 8 hours of the blood draw;
3. Patient known to be pregnant or lactating;
4. Patient with known history of bleeding diathesis or currently active bleeding;
5. Platelet count <100,000/mm the day of the blood draw;
6. Hematocrit <25% the day of the blood draw;
7. On warfarin therapy at the time of the blood draw;
8. Known blood transfusion within the preceding 10 days of the blood draw;
9. Patient who has received NSAID (not including ASA) within preceding 24 hours of the blood draw;
10. Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 patients, male or female, older than 18 years of age, who are scheduled for or underwent percutaneous coronary intervention (PCI) or CABG and have been treated with a loading dose of a thienopyridine or on a maintenance dose of a thienopyridine.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence and degree of thienopyridine resistance | Duration of hospital stay; average hospital stay of less than 48 hours
  Thienopyridine resistance will be assessed by:
  oThe VASP assay, which measures the platelet reactivity index; and/or oThe VerifyNow P2Y12 receptor inhibition assay, which measures P2Y12 reaction units (PRU); and/or oThe Chrono-Log Lumi-Aggregometer, which measures platelet aggregation (via optical density or electrical impedance) in response to ADP stimulation; and/or oThe PlaCor PRT 7000 platelet reactivity assay

SECONDARY OUTCOMES:
The prevalence of aspirin resistance | Duration of hospital stay; average hospital stay of less than 48 hours
  The prevalence and degree of aspirin resistance will be measured by the VerifyNow aspirin resistance assay.
Correlate levels of platelet reactivity with the presence of selected genetic polymorphisms | Duration of hospital stay; average hospital stay of less than 48 hours
  The presence of minor alleles in selected single nucleotide polymorphisms (SNPs) as measured by the Applied Biosystems Open Array system.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States